CLINICAL TRIAL: NCT01178177
Title: Retrospective Analysis of Radiologic Features of Invasive Pulmonary Aspergillosis in Transplant Recipients and Neutropenic Patients.Transplant Recipients and Neutropenic Patients
Brief Title: Radiologic Features of Invasive Pulmonary Aspergillosis
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Assistantant Professor, Asan Medical Center
Other Study IDs: IPA -HEM vs SOT-2010
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Hematologic Disease; Solid Organ Transplantation
Keywords: Invasive pulmonary aspergillosis; Solid organ transplantation; Hematologic disease
MeSH Terms: conditions — Hematologic Diseases; Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SOT recipients: solid organ transplant recipients with invasive pulmonary aspergillosis
- Hematologic disease: Hematologic disease patients with invasive pulmonary aspergillosis

SUMMARY:
Invasive pulmonary aspergillosis (IPA) is an opportunistic infection that primarily affects recipients of solid organ transplants (SOTs) and patients with chemotherapy- induced neutropenia.Although both of these populations are at high risk for IPA, they differ with regards to the specific defects in host defense mechanisms that increase their risk for IPA. Chemotherapy- induced neutropenia is the principal defect affecting patients with hematologic malignancies, whereas transplant recipients tend to have dysfunctional T cells and phagocytes, as a result of immunosuppressive drug therapy. Thus, the patterns of IPA-related infection and inflammation may differ according to the type of underlying immune defect. Although the clinical and radiological features of IPA in patients with neutropenia have been extensively studied, little is known about the characteristics of IPA in SOT recipients. The investigators therefore compared the IPA- related clinical and radiological findings in SOT recipients with those of neutropenic patients.

ELIGIBILITY:
Inclusion Criteria:

* IPA cases with solid organ transplant recipients and hematologic disease patients
* proven and probable invasive pulmonary aspergillosis by modified EORTC/MSG criteria

Exclusion Criteria:

* under 16 years old
* possible cases of invasive pulmonary aspergillosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients who are diagnosed with invasive pulmonary aspergillosis (IPA)between January 2008 and February 2010.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Study Chair — Department of Infectious Diseases, Asan Medical Center

REFERENCES:
- [Result] Park SY, Lim C, Lee SO, Choi SH, Kim YS, Woo JH, Song JW, Kim MY, Chae EJ, Do KH, Song KS, Seo JB, Kim SH. Computed tomography findings in invasive pulmonary aspergillosis in non-neutropenic transplant recipients and neutropenic patients, and their prognostic value. J Infect. 2011 Dec;63(6):447-56. doi: 10.1016/j.jinf.2011.08.007. Epub 2011 Aug 16. PMID 21854805